CLINICAL TRIAL: NCT06131190
Title: Effect Mindfulness Based Training on Attention, Hyperactivity and Emotion Regulation Among Children With ADHD: A Randomized Controlled Trails
Brief Title: Effect Mindfulness Training on Attention, Hyperactivity and Emotion Regulation Among Children With ADHD:
Acronym: MindADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 85-b
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-09

CONDITIONS: A
Keywords: Mindfulness; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Effect Mindfulness Based Training on Attention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): ADHD child who exposed to mindfulness training
  Interventions: Behavioral: mindfulness training
- control group (No Intervention): ADHD child take only pharmocological intervention

INTERVENTIONS:
Behavioral: mindfulness training — it focuses on attention and has gained empirical support as a complementary or alternative intervention
  Arms: study group

SUMMARY:
Mindfulness training is a promising form of training for children with ADHD, as it focuses on attention and has gained empirical support as a complementary or alternative intervention. It involves increasing awareness and nonjudgmental observation of present-moment experiences while reducing automatic responding

DETAILED DESCRIPTION:
training to sustain focus on present-moment experiences and gently shifting attention back to the meditation object when the mind drifts (Bishop, et al., 2004). Mindfulness meditation is a relatively new approach for reducing stress and emotion regulation difficulties among children. While researching the efficacy of mindfulness training in children is a new domain, existing evidence suggests that it has positive effects on psychological well-being, pain management, emotion dysregulation, negative behaviors, and cognitive/executive functions and attention (Evans et al., 2018; Zhang, Díaz-Román, & Cortese,2018).

Nurses have an important role in caring for children with ADHD, particularly in the context of mindfulness-based interventions. They can provide education and support to both parents and children regarding the benefits of mindfulness practice and can help implement mindfulness programs in clinical and community settings.

ELIGIBILITY:
Inclusion Criteria:

* age from 10-18 years old
* diagnosed with ADHD

Exclusion Criteria:

* age less than 10

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
study group | three months
  ADHD child who exposed to mindfulness training exhibit higher attention and less hyperactivity than whom not exposed (Vanderbit Assessment scale)

SECONDARY OUTCOMES:
study group | 3 monthes
  ADHD child who exposed to mindfulness training exhibit higher emotion regulationthan whom not exposed (emotional regulation inventory)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Husien, Alexandria, Please Select A Country, Egypt

REFERENCES:
- [Derived] Elzohairy NW, Elzlbany GAM, Khamis BI, El-Monshed AH, Atta MHR. Mindfulness-based training effect on attention, impulsivity, and emotional regulation among children with ADHD: The role of family engagement in randomized controlled trials. Arch Psychiatr Nurs. 2024 Dec;53:204-214. doi: 10.1016/j.apnu.2024.10.001. Epub 2024 Oct 9. PMID 39615936

DOCUMENTS (1):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT06131190/Prot_000.pdf